CLINICAL TRIAL: NCT04665739
Title: Randomized Phase II Trial of Lutetium Lu 177 Dotatate Versus Everolimus in Somatostatin Receptor Positive Bronchial Neuroendocrine Tumors
Brief Title: Testing Lutetium Lu 177 Dotatate in Patients With Somatostatin Receptor Positive Advanced Bronchial Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-12905; NCI-2020-12905 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A021901 (Other: Alliance for Clinical Trials in Oncology); A021901 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lung Neuroendocrine Tumor; Functioning Lung Neuroendocrine Tumor; Locally Advanced Lung Neuroendocrine Neoplasm; Lung Neuroendocrine Neoplasm; Lung Neuroendocrine Tumor G1; Lung Neuroendocrine Tumor G2; Metastatic Lung Neuroendocrine Neoplasm; Metastatic Lung Neuroendocrine Tumor; Non-Functioning Lung Neuroendocrine Tumor; Recurrent Lung Neuroendocrine Neoplasm; Unresectable Lung Neuroendocrine Neoplasm; Unresectable Lung Neuroendocrine Tumor
MeSH Terms: interventions — Specimen Handling; Everolimus; Fluorodeoxyglucose F18; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (lutetium Lu 177 dotatate) (Experimental): Patients receive lutetium Lu 177 dotatate IV over 30-40 minutes on day 1 of each cycle. Treatment repeats every 56 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET during screening. Patients also undergo CT or MRI during screening and on the trial as well as FDG PET and SPECT on the trial. Additionally, patients undergo blood and tissue sample collection during screening and on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography; Other: Survey Administration
- Arm II (everolimus) (Active Comparator): Patients receive everolimus PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may be able to cross-over to Arm I. Patients undergo PET during screening. Patients also undergo CT or MRI during screening and on the trial as well as FDG PET and SPECT on the trial. Additionally, patients undergo blood and tissue sample collection during screening and on the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Everolimus; Other: Fludeoxyglucose F-18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Single Photon Emission Computed Tomography; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD-001; RAD001; Votubia; Zortress
  Arms: Arm II (everolimus)
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
  Arms: Arm I (lutetium Lu 177 dotatate)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of lutetium Lu 177 dotatate compared to the usual treatment (everolimus) in treating patients with somatostatin receptor positive bronchial neuroendocrine tumors that have spread to other places in the body (advanced). Lutetium Lu 177-dotate is a radioactive drug. It binds to a protein called somatostatin receptor, which is found on some neuroendocrine tumor cells. Lutetium Lu 177-dotatate builds up in these cells and gives off radiation that may kill them. It is a type of radioconjugate and a type of somatostatin analog. Lutetium Lu 177 dotatate may be more effective than everolimus in shrinking or stabilizing advanced bronchial neuroendocrine tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) of receiving lutetium Lu 177 dotatate to that of receiving everolimus in patients with bronchial neuroendocrine tumor (NET).

SECONDARY OBJECTIVES:

I. To compare the overall survival (OS) of receiving lutetium Lu 177 dotatate versus everolimus in patients with bronchial NET.

II. To compare the overall response rate (ORR) associated with lutetium Lu 177 dotatate versus everolimus in patients with bronchial NET.

III. To evaluate and compare the toxicity profile of lutetium Lu 177 dotatate and everolimus.

EXPLORATORY OBJECTIVES:

I. To study late toxicities of lutetium Lu 177 dotatate therapy including renal dysfunction, myelodysplastic syndrome, and acute leukemia.

II. To study the impact of pretreatment disease burden, somatostatin receptor status on lutetium Lu 177 dotatate (DOTATATE) positron emission tomography (PET) (or other somatostatin receptor [SSTR]-PET), and measured dosimetry of response.

III. To evaluate the response rate (RR) and other efficacy parameters in typical and atypical carcinoid based on central retrospective pathology review.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive lutetium Lu 177 dotatate intravenously (IV) over 30-40 minutes on day 1 of each cycle. Treatment repeats every 56 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PET during screening. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on the trial as well as fludeoxyglucose F-18 (FDG) PET and single photon emission computed tomography (SPECT) on the trial. Additionally, patients undergo blood and tissue sample collection during screening and on the trial.

ARM II: Patients receive everolimus orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression may be able to cross-over to Arm I. Patients undergo PET during screening. Patients also undergo CT or MRI during screening and on the trial as well as FDG PET and SPECT on the trial. Additionally, patients undergo blood and tissue sample collection during screening and on the trial.

After completion of study treatment, patients are followed up every 3 months until disease progression and then every 6 months for up to 5 years following study registration.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION: Pathologic Documentation: Well- or moderately-differentiated neuroendocrine tumor(s) of bronchial origin (i.e. carcinoid) as assessed by local pathology

  * The pathology report must state ONE of the following:

    * Well- or moderately-differentiated neuroendocrine tumor,
    * Low- or intermediate-grade neuroendocrine tumor, or
    * Carcinoid tumor (including typical or atypical carcinoid tumors)
* PRE-REGISTRATION: Documentation of histology from a primary or metastatic site is allowed
* PRE-REGISTRATION: Functional (evidence of peptide hormones and/or bioactive substances associated with a clinical hormone syndrome such as carcinoid syndrome or Cushing's syndrome) or nonfunctional tumors are allowed
* PRE-REGISTRATION: Patients with poorly-differentiated or high-grade neuroendocrine carcinoma (i.e. large cell neuroendocrine carcinoma of lung, small cell lung cancer) or mixed tumors (i.e. adenocarcinoid tumor) are not eligible
* PRE-REGISTRATION: Recurrent or locally-advanced/unresectable or metastatic disease
* PRE-REGISTRATION: Neuroendocrine tumor of bronchial (i.e. lung) primary site
* PRE-REGISTRATION: Lesions must have shown radiological evidence of disease progression in the 12 months prior to pre-registration

  * Tumor must have shown somatostatin receptor (SSTR) positivity on 68Ga-DOTATATE PET or other SSTR-PET scan in the 12 months prior to pre-registration; however, documentation of SSTR positivity in the 6 months prior to pre-registration is preferred. SSTR positivity is defined as uptake greater than background liver in all measurable lesions
* PRE-REGISTRATION: Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 by computer tomography (CT) scan or magnetic imaging (MRI). Any lesions which have undergone percutaneous therapies or radiotherapy should not be considered measurable unless the lesion has clearly progressed since the procedure
* PRE-REGISTRATION: Lesions must be accurately measured in at least one dimension (longest diameter to be recorded) as >= 1 cm with CT or MRI (or >= 1.5 cm short axis for lymph nodes). Non-measurable disease includes disease smaller than these dimensions or lesions considered truly non-measurable including: leptomeningeal disease, bone metastases, ascites, pleural or pericardial effusion, lymphangitic involvement of skin or lung
* REGISTRATION: Confirmation of SSTR positivity by Alliance Imaging Core Lab (ICL) at Imaging and Radiation Oncology Core (IROC) Ohio central radiographic review
* REGISTRATION: Patients with treatment-naive or previously-treated disease are allowed. Patients with previously-treated disease must have demonstrated radiographic disease progression on the prior therapy
* REGISTRATION: No prior treatment with peptide receptor radionuclide therapy (PRRT) (e.g. lutetium Lu 177 dotatate)
* REGISTRATION: No prior treatment with mammalian target of rapamycin (mTOR) inhibitors (e.g. deforolimus, everolimus, sirolimus, temsirolimus, etc.)
* REGISTRATION: Prior treatment with hepatic artery embolization (including bland embolization, chemoembolization, and selective radioembolization) or ablative therapies (i.e. cryoablation, radiofrequency ablation, etc.) is allowed if measurable disease remains outside of the treated area or if there is documented disease progression in a treated site. Prior liver-directed (including ablative) treatment must be completed at least 28 days prior to registration
* REGISTRATION: Prior treatment with 90-Yttrium radioembolization must be completed at least 6-weeks prior to registration
* REGISTRATION: Radiation therapy to the lung and/or mediastinum must be completed at least 14 days prior to registration for stereotactic ablative and at least 28 days prior to registration for conventional fractionation
* REGISTRATION: Prior treatment with systemic anticancer therapy must be completed at least 28 days prior to registration (except for somatostatin analogs in patients with functional tumors). Continuation of treatment with somatostatin analogs while on protocol therapy is allowed provided that the patient:

  * Has functional tumors (evidence of peptide hormones and/or bioactive substances associated with a clinical hormone syndrome such as carcinoid syndrome or Cushing's syndrome), and
  * Has previously demonstrated radiographic disease progression while on somatostatin analog therapy
* REGISTRATION: Patients must have completed any major surgery at least 28 days prior to registration. Complete wound healing from major surgery should occur prior to registration
* REGISTRATION: Patients should have improvement of any toxic effects of prior therapy (except alopecia, fatigue, and other non-reversible toxic effects such as neuropathy from cisplatin) to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, grade 1 or less
* REGISTRATION: Not pregnant and not nursing

  * Therefore, for women of childbearing potential only, a negative pregnancy test done =< 28 days prior to registration is required
* REGISTRATION: Age >= 18 years
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* REGISTRATION: Hemoglobin >= 8.0 g/dL
* REGISTRATION: Platelet count >= 75,000/mm^3
* REGISTRATION: Absolute neutrophil count (ANC) >= 1,500/mm^3
* REGISTRATION: Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance >= 40 mL/min

  * Calculated by the Cockcroft-Gault equation
* REGISTRATION: Total bilirubin =< 2.0 x ULN

  * In patients with Gilbert's syndrome, if total bilirubin is > 2.0 x ULN, then direct bilirubin must be =< 2.0 x ULN
* REGISTRATION: Albumin >= 2.8 g/dL
* REGISTRATION: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3.0 x ULN
* REGISTRATION: No known central nervous system metastases unless treated and clinically stable for at least 14 days prior to registration. Patients on steroid support must be clinically stable on weaning doses of steroids
* REGISTRATION: No other currently active malignancy that requires therapy or is expected to require therapy during the study (excluding non-melanoma skin cancers or in situ carcinomas, such as breast or cervical)
* REGISTRATION: No known active hepatitis B (defined as hepatitis B surface antigen [HbsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] viral load detected). The exception is for patients with known active hepatitis B virus (defined as HbsAg reactive) infection, where the HBV viral load must be undetectable on suppressive therapy for patient to be eligible
* REGISTRATION: Patients with known human immunodeficiency virus (HIV) infections on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* REGISTRATION: No known active or uncontrolled infections requiring ongoing antifungals or antibiotics in the 3 days prior to registration
* REGISTRATION: No receipt of live attenuated vaccines in the 7 days prior to registration
* REGISTRATION: No known decompensated liver cirrhosis
* REGISTRATION: No known prior drug-induced pneumonitis that was symptomatic or required treatment
* REGISTRATION: No known medical condition causing an inability to swallow and no known impairment of gastrointestinal function that may significantly alter the absorption of an oral agent
* REGISTRATION: No known hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus, etc.)
* REGISTRATION: Concurrent somatostatin analog use while on protocol therapy is allowed provided that the patient: 1) has a functional tumor (evidence of peptide hormones and/or bioactive substances associated with a clinical hormone syndrome such as carcinoid syndrome or Cushing's syndrome), 2) has previously demonstrated radiographic disease progression while on somatostatin analog therapy
* REGISTRATION: Chronic concomitant treatment with P-gp and strong CYP3A4 inhibitors and/or inducers is not allowed on the everolimus treatment arm of this study. Given that the study is randomized, all patients on P-gp and strong CYP3A4 inhibitors and/or inducers must discontinue the drug(s) 7 days prior to registration
* RE-REGISTRATION: Confirmation of disease progression by RECIST v1.1 by real-time Alliance ICL at IROC Ohio central radiographic review
* RE-REGISTRATION: Not pregnant and not nursing

  * Women of childbearing potential only, a negative pregnancy test done =< 28 days prior to re-registration is required
* RE-REGISTRATION: ECOG performance status 0-2
* RE-REGISTRATION: Hemoglobin >= 8.0 g/dL
* RE-REGISTRATION: Platelet count >= 75,000/mm^3
* RE-REGISTRATION: Absolute neutrophil count (ANC) >= 1,500/mm^3
* RE-REGISTRATION: Creatinine =< 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance >= 40 mL/min

  * Calculated by the Cockcroft-Gault equation
* RE-REGISTRATION: Total bilirubin =< 2.0 x ULN

  * In patients with Gilbert's syndrome, if total bilirubin is > 2.0 x ULN, then direct bilirubin must be =< 2.0 x ULN
* RE-REGISTRATION: Albumin >= 2.8 g/dL
* RE-REGISTRATION: AST/ALT =< 3.0 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2033-01-16 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival (PFS) | From randomization until either radiographic progression confirmed by central radiology review or death, assessed up to 5 years from study registration
  Will be compared between patients with a bronchial neuroendocrine tumor receiving lutetium Lu 177 dotatate to those receiving everolimus. The distribution of PFS will be estimated using the Kaplan Meier method. Will be tested using a one-sided stratified log rank test. The median PFS, along with 90% confidence intervals (CIs), will be estimated for the two treatment groups.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until death due to any cause, with patients censored at the last date known to be alive or last contact date, assessed up to 5 years from study registration
  The distribution of OS will be estimated using the method of Kaplan-Meier. The median OS, along with 90% CIs, will be estimated by the two treatment groups. OS will be compared between the two between treatment arms using the stratified log-rank test at a one-sided 10% level of significance.
Overall response rate (ORR) | Up to 5 years from study registration
  Defined as the proportion of patients in each arm whose best response is either complete response (CR) or partial response (PR). Will be estimated using point estimates and 95% CIs according to the methods in Duffy and Santner.
Incidence of adverse events | Up to 5 years from study registration
  Will evaluate and compare the toxicity profile of lutetium Lu 177 dotatate and everolimus. As per National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0, the term toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to the study treatment.

OTHER OUTCOMES:
Incidence of late toxicities of lutetium Lu 177 dotatate therapy | More than 30 days after treatment
  The incidence of grade 3+ late toxicities will be analyzed in a descriptive manner. Incidence will be described for each treatment arm. Frequency tables will be reviewed for patterns.
Pretreatment disease burden | Baseline
Somatostatin receptor (SSTR) status on DOTATATE positron emission tomography (PET) (or other SSTR-PET) | Up to 5 years from study registration
Dosimetry of response | Up to 5 years from study registration
Response rate | Up to 5 years from study registration
  The proportion of patients in each carcinoid group with either CR or PR as their best response will be estimated using point estimates and 95% CIs according to the methods in Duffy and Santner. ORR will be compared between treatment arms using the 2-sample z-test to compare sample proportion at a one-sided 5% level of significance.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (29):
- United States (29):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm